CLINICAL TRIAL: NCT02740374
Title: A Prospective, Randomized, Parallel-group Single Center Study to Evaluate the Use of Thromboelastometry (ROTEM) in Patients Undergoing Spine Surgeries
Brief Title: Evaluation of Thromboelastometry (ROTEM) During Spinal Surgery
Acronym: ROTEM_SPINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Galina Dimitrova, M.D, Principal INvestigator, Clinical Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014H0447
Record Dates: First submitted 2016-01-05; First posted 2016-04-15 (Estimated); Results first posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Blood Loss, Surgical
Keywords: ROTEM; Thromboelastometry; spine surgery; allogenic blood transfusion; blood loss; red blood cell transfusion
MeSH Terms: conditions — Blood Loss, Surgical; Hemorrhage | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ROTEM (Experimental): ROTEM will be performed in patients with signs of clinically relevant bleeding and in whom blood transfusion is considered (Temp above 35 Celsius degrees; pH below 7.2; Cai above 4.6 mg/dL; Hb below 9g/dL, or below 10g/dL with anticipated greater blood loss) or at a fixed range every 2 hours or at Anesthesiologist criteria based on patient's clinical situation.
  There will be also be performed standard of care test for this set of patients, as described for the CONTROL arm. ROTEM results will guide transfusion strategy.
  Interventions: Device: ROTEM
- CONTROL/STANDARD OF CARE (Active Comparator): If patients are randomized to standard coagulation tests (SCT), these will be performed according to Ohio State Wexner University Medical Center standard practices and attending's criteria, or at 2 hour intervals per protocol.
  Standard of care tests include but are not limited to: hemoglobin, platelet count, fibrinogen concentration, INR, aPTT, and PT. These will be performed at fixed time points (preoperatively, every 2 hours intraoperatively, procedure completion, and 24 hours after procedure completion). Arterial blood gases will be performed repetitively intraoperatively at a fixed range every 1-hour or at attending's criteria, as well as any postoperative laboratory tests. SCT will guide transfusion management.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: ROTEM — ROTEM coagulation assessment and guided transfusion management.
  Arms: ROTEM
Other: Standard of Care — Standard Coagulation Tests assessment and guided transfusion management
  Arms: CONTROL/STANDARD OF CARE

SUMMARY:
The purpose of this study is to determine whether the use of ROTEM, during spinal surgery is effective on diminishing the total blood loss and the risk of Allogenic Transfusion of Blood Products vs control cases without ROTEM assessment.

DETAILED DESCRIPTION:
Study methods This is a prospective, randomized parallel-group single center study in patients undergoing elective major spine surgery. Patients will be randomized to ROTEM-guided hemostatic therapy algorithm or standard of care hemostatic therapy: arterial blood gas analysis (ABG), normalized index ratio (INR), prothrombin time (PT), thromboplastin time (aPTT), hemoglobin (Hb), platelets, and fibrinogen.

Study Procedures Patients will be randomized in a 1:1 ratio to either standard of care coagulation tests (SOC) or ROTEM. No changes in surgery or anesthesia technique will be made for the purposes of the study.

Standard of Care Coagulation Tests If patients are randomized to standard of care coagulation tests, these will be performed according to Ohio State University Wexner Medical Center standard practices and attending's criteria.

Standard of care tests include but are not limited to: hemoglobin, platelet count, fibrinogen concentration, INR, aPTT, and PT. These will be performed at fixed time points (preoperatively, every 2 hours intraoperatively, procedure completion, and 24 hours after procedure completion). Arterial blood gases will be performed repetitively intraoperative at a fixed range every 1-hour or at attending's criteria, as well as any postoperative laboratory tests.

ROTEM If patients are randomized to ROTEM, the anesthesiologist will be blinded to any intraoperative conventional coagulation test that might be performed.

ROTEM will be used according to the manufacturer's instructions, using equipment and test reagents provided by Tem International GmbH. All tests will be performed at the bedside by a clinical perfusionist trained to perform ROTEM. A specific algorithm has been created and should be followed according to clinical criteria

ROTEM monitoring will be performed in patients with signs of clinically relevant diffuse bleeding and in whom blood transfusion is considered (Temp >35 Celsius degrees; pH lower than 7.2; Cai above 4.6 mg/dL; Hb below 9g/dL, or below 10g/dL with anticipated greater blood loss) or at a fixed range every 2 hours or at Anesthesiologist criteria based on patient's clinical situation.

Patient´s clinical situation should be consider as the most important component on the transfusion decision-making process. Packed erythrocytes will be transfused to maintain hemoglobin concentrations higher 9g/dl and higher 10g/dl in individuals with underlying cardiovascular disease or anticipated greater blood loss. Individual based dynamics strongly indicating the need for erythrocyte transfusion at anesthesiologist criteria will be also part of the transfusion making decision-making process (tachycardia, hypotension, sings of ischemia on electrocardiogram, lactic acidosis, and dynamics of bleeding).

Assessment and reporting of Adverse Events The occurrence of adverse events (AE) and serious adverse events (SAE) will be recorded from the time of consent until discharge. For each AE, the relationship to the study procedures and monitoring, severity, expectedness, outcome will be determined by the PI and recorded in the study source accordingly If the case a subject withdraws from the study due to a serious adverse event the local Institutional Review Board (IRB) will be notified within 10 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18 years or older.
2. Able to provide inform consent or have a legal authorized representative able to sign consent on the patients behalf.
3. Female subject with a negative urine or serum pregnancy test, or not of childbearing potential, defined as surgically sterile due to bilateral tubal ligation, bilateral oophorectomy or hysterectomy; or are postmenopausal for at least 1 year.
4. Patients schedule to undergo elective neurosurgery, orthopedic, or combined procedures that are expected to receive blood products intraoperatively.

   -

Exclusion Criteria:

1. Subjects younger than 18 years old.
2. Subjects who are prisoners.
3. Subjects who refuse transfusion of blood products.
4. Females who are pregnant or breastfeeding.
5. Subjects unable to participate in the study for any reason in the opinion of the Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-11; Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galina Dimitrova, MD, Principal Investigator — Ohio State University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ROTEM: ROTEM will be performed in patients with signs of clinically relevant bleeding and in whom blood transfusion is considered (Temp above 35 Celsius degrees; pH below 7.2; Cai above 4.6 mg/dL; Hb below 9g/dL, or below 10g/dL with anticipated greater blood loss) or at a fixed range every 2 hours or at Anesthesiologist criteria based on patient's clinical situation.
  There will be also be performed standard of care test for this set of patients, as described for the CONTROL arm. ROTEM results will guide transfusion strategy.
  ROTEM: ROTEM coagulation assessment and guided transfusion management.
- CONTROL/STANDARD OF CARE: If patients are randomized to standard coagulation tests (SCT), these will be performed according to Ohio State Wexner University Medical Center standard practices and attending's criteria, or at 2 hour intervals per protocol.
  Standard of care tests include but are not limited to: hemoglobin, platelet count, fibrinogen concentration, INR, aPTT, and PT. These will be performed at fixed time points (preoperatively, every 2 hours intraoperatively, procedure completion, and 24 hours after procedure completion). Arterial blood gases will be performed repetitively intraoperatively at a fixed range every 1-hour or at attending's criteria, as well as any postoperative laboratory tests. SCT will guide transfusion management.
  Standard of Care: Standard Coagulation Tests assessment and guided transfusion management
Period: Overall Study
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Started | 55 | 57
Completed | 55 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE | Total
Number analyzed (Participants) | 55 | 57 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 57 | 112
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.84 (12.84) | 61.32 (11.03) | 60.1 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 29 | 65
  Male | 19 | 28 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 54 | 55 | 109
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 54 | 54 | 108
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 55 | 57 | 112

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Needing an Intraoperative Autologue Blood Product Transfusion
Description: Intraoperative Autologue Blood Product Transfusion
Time Frame: Within surgery
Population: Red blood cell
Measure: Count of Participants; unit: Participants
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
Participants | 24 | 24

2. Secondary Outcome: Postoperative Blood Product Transfusion
Description: Fresh frozen plasma transfusion.
Time Frame: Within postoperative 24 hours
Population: Fresh frozen plasma transfusion.
Measure: Count of Participants; unit: Participants
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
Participants | 1 | 3

3. Secondary Outcome: Number of Participants Requiring Cryoprecipitate Transfusion
Description: Number of participants
Time Frame: Perioperative- up to 24 hours after surgery start time (cumulative)
Population: Cryoprecipitate Transfusion Requirements
Measure: Count of Participants; unit: Participants
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
Participants | 1 | 2

4. Secondary Outcome: Number of Participants Requiring Platelet Transfusion
Description: Number of participants
Time Frame: Perioperative- up to 24 hours after surgery start time (cumulative)
Population: Platelet Transfusion Requirements
Measure: Count of Participants; unit: Participants
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
Participants | 1 | 6

5. Secondary Outcome: Fibrinogen Concentrate Transfusion Requirements
Description: Percentage
Time Frame: Within Surgery and Postoperative 24 hours
Population: Fibrinogen concentrate Transfusion Requirements
Measure: Count of Participants; unit: Participants
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
Participants | 0 | 0

6. Secondary Outcome: Prothrombin Complex Transfusion Requirements
Description: Percentage
Time Frame: Within Surgery and Postoperative 24 hours
Population: Prothrombin Complex transfusion Requirements
Measure: Count of Participants; unit: Participants
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
Participants | 0 | 0

7. Secondary Outcome: Factor VII Transfusion Requirements
Description: Percentage
Time Frame: Within Surgery and Postoperative 24 hours
Population: Factor VII Transfusion Requirements
Measure: Count of Participants; unit: Participants
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
Participants | 0 | 0

8. Secondary Outcome: Need for Mechanical Ventilation During Postoperative Period
Time Frame: Within 30 days after surgery
Population: Need for mechanical Ventilation During Postoperative period
Measure: Count of Participants; unit: Participants
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
Participants | 8 | 3

9. Secondary Outcome: Length of Stay on Intensive Care Unit (ICU)
Time Frame: Within 30 days after surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
minutes | 3952.38 (3304.78) | 4915.85 (3298.3)

10. Secondary Outcome: Length of Stay on Post Anesthesia Care Unit (PACU)
Time Frame: Within 30 days after surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
minutes | 183.03 (189.27) | 171.81 (200.48)

11. Secondary Outcome: Overall Hospital Stay
Time Frame: Within 30 days after surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
minutes | 8535.49 (4656.84) | 1095.61 (7617.49)

12. Secondary Outcome: Surgical Site Infection
Time Frame: within 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
Participants | 3 | 6

13. Secondary Outcome: Mortality
Description: 30 day mortality
Time Frame: within 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
Participants | 1 | 1

14. Secondary Outcome: Cardiovascular Complications Rate
Time Frame: within Postoperative 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
Participants | 2 | 0

15. Secondary Outcome: Thromboembolic Complications Rate
Time Frame: within Postoperative 30 days
Population: Thromboembolic Complications rate
Measure: Count of Participants; unit: Participants
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
Participants | 0 | 2

16. Secondary Outcome: Respiratory Complications Rate
Time Frame: Within postoperative 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
Participants | 3 | 4

17. Secondary Outcome: Renal System Complications Rate
Time Frame: Within 30 postoperative days
Measure: Count of Participants; unit: Participants
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
Participants | 1 | 2

18. Secondary Outcome: Cerebrovascular Complications Rate
Time Frame: within 30 postoperative days
Measure: Count of Participants; unit: Participants
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
Participants | 0 | 1

19. Secondary Outcome: Infectious Complications Rate
Time Frame: Within postoperative 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
Participants | 1 | 5

20. Secondary Outcome: Reintervention Related to Postoperative Bleeding Rate
Time Frame: Within postoperative 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
Number analyzed (Participants) | 55 | 57
Participants | 5 | 2

21. Other Pre Specified Outcome: Cost Comparison
Description: Compare costs of ROTEM guided therapy or Standard of Care guided therapy.
Time Frame: within 30 days after surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | ROTEM | CONTROL/STANDARD OF CARE
All-Cause Mortality (participants affected / at risk) | 1/55 | 1/57
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/57
Other Adverse Events (participants affected / at risk) | 0/55 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-04-21): https://cdn.clinicaltrials.gov/large-docs/74/NCT02740374/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT02740374/ICF_001.pdf